CLINICAL TRIAL: NCT00664560
Title: Randomized, Double-Blind, Parallel Group, Placebo-Controlled Multi-Center Study Evaluating the Efficacy of PN400 (VIMOVO) Twice Daily (Bid) and Celecoxib Once Daily (qd) in Patients With Osteoarthritis of the Knee
Brief Title: Efficacy Study of PN400 (VIMOVO) Twice Daily and Celebrex Once Daily in Patients With Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: POZEN (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PN400-307
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARM 1 PN 400 (VIMOVO) (Experimental): PN400: 500 mg naproxen/20 mg esomeprazole
  Interventions: Drug: PN 400 (VIMOVO); Drug: Rescue Antacid
- Arm 2 (celebrex) (Active Comparator): Celecoxib 200 mg
  Interventions: Drug: celebrex; Drug: Rescue Antacid
- Arm 3 (placebo) (Placebo Comparator): sugar pill
  Interventions: Drug: Placebo; Drug: Rescue Antacid

INTERVENTIONS:
Drug: PN 400 (VIMOVO) — 500 mg naproxen/20 mg esomeprazole bid
  Other Names: PN 400
  Arms: ARM 1 PN 400 (VIMOVO)
Drug: celebrex — 200 mg celecoxib qd
  Arms: Arm 2 (celebrex)
Drug: Placebo — sugar pill bid
  Arms: Arm 3 (placebo)
Drug: Rescue Antacid — Antacid Tablets

SUMMARY:
We will evaluate the efficacy of PN400 and an active comparator in patients that have Osteoarthritis of the knee.

DETAILED DESCRIPTION:
3-Month study in subjects 50 years and older with osteoarthritis of the knee. Assessments Western Ontario and McMaster Universities (WOMAC) pain and function and patient global assessment scales.

ELIGIBILITY:
Inclusion Criteria

1. Male or non-pregnant female subjects50 years of age and older with a 6-month history of OA of the knee
2. Female subjects were eligible for participation in the study if they were of non-childbearing potential (i.e., physiologically incapable of becoming pregnant); or of childbearing potential, had a negative pregnancy test at Screening, and using adequate contraceptive methods.
3. Subjects were required to have been on a stable dose of NSAIDs, COX-2 inhibitors or other oral analgesic therapy for at least 6 weeks and required to continue treatment for 12 weeks. Current oral analgesic therapy was withdrawn at Screening.
4. Each subject was required to be able to understand and comply with study procedures required of a subject and was able and willing to provide written informed consent prior to any study procedures being performed.
5. Subjects were required to agree to keep physical activity at a stable level throughout the study.
6. Subjects were required to have symptomatic OA of the knee meeting American College of Rheumatology (ACR) criteria for clinical diagnosis of OA.
7. Subjects were required to have an ACR functional class rating of I, II or III. In addition, subjects meet the requirements for OA flare at the Baseline/ Randomization Visit.

Exclusion Criteria

1. Subjects with rheumatoid arthritis or gout/pseudo-gout
2. Subjects with fibromyalgia syndrome
3. Acute joint trauma at the index joint within the 3 months prior to screen with active symptoms
4. Previous (in the past 12 months) or anticipated need for surgical or invasive procedure performed on the index joint during the study
5. Subject was currently taking or anticipated to take Coumadin®, warfarin, or lithium
6. History of hypersensitivity to esomeprazole or to another PPI
7. History of allergic reaction or intolerance to any NSAID (including aspirin) and/or subject had a history of NSAID-induced symptoms of asthma, rhinitis, and/or nasal polyps
8. History of allergic reactions to sulfonamides
9. Subjects with intra-articular or intramuscular corticosteroids or intra-articular hyaluronic acid injections within 8 weeks prior to randomization
10. Participation in any study of an investigational treatment in the 4 weeks before Screening
11. Presence of uncontrolled acute or chronic medical illness, e.g. morbid obesity, GI disorder, diabetes, active GI disease, chronic or acute renal or hepatic disorder, depression and/or infection, etc, that would endanger a subject if the subject were to participate in the study
12. GI disorder (e.g., severe erosive esophagitis, Zollinger Ellison syndrome) or surgery leading to impaired drug absorption
13. Peptic ulcer disease within 6 months prior to Screening
14. Evidence of uncontrolled, or unstable cardio- or cerebrovascular disorder, which in the investigator's opinion would have endangered a subject if the subject were to participate in the study
15. Schizophrenia or bipolar disorder
16. Subjects who had started physical therapy on the index joint less than 6 weeks prior to study Screening
17. Use of any excluded concomitant medication
18. A recent history (in the past 3 months) suggestive of alcohol or drug abuse or dependence, including overuse/abuse of narcotics for management of pain
19. Serious blood coagulation disorder including use of systemic anti-coagulants
20. Screening laboratory value for alanine aminotransferase, aspartate aminotransferase greater than 2 times the upper limit of normal
21. Estimated creatinine clearance less than 30 ml/min
22. Other than noted specifically, any Screening laboratory value that was clinically significant in the investigator's opinion and would have endangered a subject if the subjects were to participate in the study
23. History of malignancy, treated or untreated, within the past 5 years, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin
24. Previous participation in another PN 400 clinical research trial
25. Subjects who were employees of the research facility or who were in some way under the supervision of the principal investigator for this study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everardus Orlemans, PhD, Study Chair — POZEN
Locations (1):
- POZEN, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Holt RJ, Fort JG, Grahn AY, Kent JD, Bello AE. Onset and durability of pain relief in knee osteoarthritis: Pooled results from two placebo trials of naproxen/esomeprazole combination and celecoxib. Phys Sportsmed. 2015 Jul;43(3):200-12. doi: 10.1080/00913847.2015.1074852. Epub 2015 Aug 3. PMID 26313454
- [Derived] Holt RJ, Fort JG, Grahn AY, Kent JD, Bello AE. Onset and durability of pain relief in knee osteoarthritis: pooled results from two placebo trials of naproxen/esomeprazole combination and celecoxib. Phys Sportsmed. 2015 Aug 3:1-13. Online ahead of print. PMID 26235613
- [Derived] Hochberg MC, Fort JG, Svensson O, Hwang C, Sostek M. Fixed-dose combination of enteric-coated naproxen and immediate-release esomeprazole has comparable efficacy to celecoxib for knee osteoarthritis: two randomized trials. Curr Med Res Opin. 2011 Jun;27(6):1243-53. doi: 10.1185/03007995.2011.580340. Epub 2011 Apr 28. PMID 21524238

RESULTS

PARTICIPANT FLOW:
Groups:
- (PN 400 (VIMOVO) Twice Daily): PN 400 (VIMOVO): 500 mg naproxen/20 mg esomeprazole
- (Celebrex 200 mg Once Daily): Celecoxib 200 mg (Celebrex) taken once daily
- (Placebo Twice Daily): placebo (sugar pill) dosed twice daily (bid)
Period: Overall Study
Arm/Group | (PN 400 (VIMOVO) Twice Daily) | (Celebrex 200 mg Once Daily) | (Placebo Twice Daily)
Started | 247 (Safety Population) | 243 (Safety Population) | 124 (Safety Population)
Completed | 208 | 208 | 105
Not Completed | 39 | 35 | 19
Not completed — Adverse Event | 19 | 16 | 7
Not completed — Withdrawal by Subject | 9 | 13 | 7
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Other | 11 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | (PN 400 (VIMOVO) Twice Daily) | (Celebrex 200 mg Once Daily) | (Placebo Twice Daily) | Total
Number analyzed (Participants) | 247 | 243 | 124 | 614
Age Continuous [Mean (Standard Deviation); unit: years] | 62.5 (7.7) | 61.5 (8.0) | 61.6 (8.2) | 61.9 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 148 | 82 | 392
  Male | 85 | 95 | 42 | 222

OUTCOME MEASURES:

1. Primary Outcome: Change in Western Ontario and McMaster Universities (WOMAC) Pain Questionnaire Subscore From Baseline
Description: Western Ontario and McMaster Universities (WOMAC) pain questionnaire has 5 questions on pain all use visual analog scale (VAS) of 100 mm, with 0 mm being "no pain" and 100 mm being "extreme pain". The outcome measures a change in WOMAC pain at 12 weeks from baseline (in mm). WOMAC is a self-administered, patient-reported health status questionnaire designed to capture elements of pain, stiffness and physical disability in patients with OA of the knee and/or hip joints. It consists of 24 questions (5 questions about pain, 2 on stiffness and 17 about physical function).
Time Frame: Baseline and 12 weeks
Population: Analysis Population: Baseline + took >= 1 dose + >= 1 post-baseline WOMAC efficacy evaluation (intent-to-treat population). Used Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | (PN 400 (VIMOVO) Twice Daily) | (Celebrex 200 mg Once Daily) | (Placebo Twice Daily)
Number analyzed (Participants) | 226 | 221 | 108
mm | -43.4 (26.8) | -41.1 (26.2) | -34.0 (25.3)
Statistical Analysis 1: Comparison: (PN 400 (VIMOVO) Twice Daily) vs (Celebrex 200 mg Once Daily); Test type: Non-Inferiority or Equivalence — Non-Inferiority (NI) margin of 10mm between Arm 1 and Arm 2 (NI design uses confidence intervals, not p-values); ANCOVA; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-4.76 to 4.32]

2. Primary Outcome: Change in Western Ontario and McMaster Universities (WOMAC) Function Questionnaire Subscore From Baseline
Description: WOMAC function questionnaire (VAS). The 17 questions about function all use visual analog scale (VAS) of 100 mm; 0 mm being "no pain" and 100 mm being "extreme pain". The outcome measures a change in WOMAC pain from baseline (in mm).
  The Western Ontario and McMaster Universities (WOMAC) is a self-administered, patient-reported health status questionnaire that is designed to capture elements of pain, stiffness and physical disability in patients with OA of the knee and/or hip joints. The index consists of 24 questions (5 questions about pain, 2 on stiffness and 17 about physical function).
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | (PN 400 (VIMOVO) Twice Daily) | (Celebrex 200 mg Once Daily) | (Placebo Twice Daily)
Number analyzed (Participants) | 226 | 221 | 108
mm | -37.5 (27.1) | -36.0 (26.4) | -28.9 (24.9)
Statistical Analysis 1: Comparison: (PN 400 (VIMOVO) Twice Daily) vs (Celebrex 200 mg Once Daily); Test type: Non-Inferiority or Equivalence — 10 mm Non-Inferiority (NI) margin between Arm 1 and Arm 2 (NI design uses confidence intervals, not p-values); ANCOVA; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-4.57 to 4.38]

3. Primary Outcome: Change in Patient Global Assessment (PGA) Subscore From Baseline
Description: PGA questionnaire. The patient global assessment (PGA) question asks about how the subject is doing considering his/her arthritis and is measured by a visual analog scale (VAS); 0 mm (very poor) 100 mm (excellent). The outcome measures a change from baseline PGA in mm.
Time Frame: 12 weeks
Population: Analysis Population: Baseline + took >= 1 dose + >= 1 post-baseline PGA efficacy evaluation (intent-to-treat population). Used Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | (PN 400 (VIMOVO) Twice Daily) | (Celebrex 200 mg Once Daily) | (Placebo Twice Daily)
Number analyzed (Participants) | 242 | 230 | 119
mm | 21.5 (33.4) | 22.4 (28.7) | 12.4 (28.9)
Statistical Analysis 1: Comparison: (PN 400 (VIMOVO) Twice Daily) vs (Celebrex 200 mg Once Daily); Test type: Non-Inferiority or Equivalence — Non-Inferiority (NI) margin 10 mm between Arm 1 and Arm 2 (NI design uses confidence intervals, not p-values); ANCOVA; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-5.08 to 4.14]

4. Secondary Outcome: American Pain Society Patient Outcome Questionnaire (APS-POQ)Total Interference Caused by Pain.
Description: Mean change from Baseline scores calculated for each subject through Day 7. Scale 0 through 70, where 0=no pain interference and 70=complete interference.
Time Frame: Baseline and Day 7
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | (PN 400 (VIMOVO) Twice Daily) | (Celebrex 200 mg Once Daily) | (Placebo Twice Daily)
Number analyzed (Participants) | 246 | 242 | 124
Units on a scale | -17.8 (14.3) | -17.7 (16.0) | -12.8 (13.6)

5. Secondary Outcome: Change in Western Ontario and McMaster Universities (WOMAC) Pain Questionnaire Subscore From Baseline
Description: Western Ontario and McMaster Universities (WOMAC) pain questionnaire has 5 questions on pain all use visual analog scale (VAS) of 100 mm, with 0 mm being "no pain" and 100 mm being "extreme pain". The outcome measures a change in WOMAC pain at 6 weeks from baseline (in mm). WOMAC is a self-administered, patient-reported health status questionnaire designed to capture elements of pain, stiffness and physical disability in patients with OA of the knee and/or hip joints. It consists of 24 questions (5 questions about pain, 2 on stiffness and 17 about physical function).
Time Frame: Week 6
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | (PN 400 (VIMOVO) Twice Daily) | (Celebrex 200 mg Once Daily) | (Placebo Twice Daily)
Number analyzed (Participants) | 198 | 187 | 101
mm | -40.9 (26.9) | -39.4 (25.4) | -30.7 (25.5)

6. Secondary Outcome: Change in Western Ontario and McMaster Universities (WOMAC) Function Questionnaire Subscore From Baseline
Description: as for outcome 2
Time Frame: Week 6
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | (PN 400 (VIMOVO) Twice Daily) | (Celebrex 200 mg Once Daily) | (Placebo Twice Daily)
Number analyzed (Participants) | 198 | 187 | 101
mm | -35.3 (26.9) | -33.9 (25.6) | -27.3 (26)

7. Secondary Outcome: Change in Patient Global Assessment (PGA) Subscore From Baseline
Description: as for outcome 3
Time Frame: Week 6
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | (PN 400 (VIMOVO) Twice Daily) | (Celebrex 200 mg Once Daily) | (Placebo Twice Daily)
Number analyzed (Participants) | 239 | 227 | 119
mm | 22.6 (31.6) | 20.7 (28.8) | 14.7 (29.3)

8. Secondary Outcome: Antacid Tablet Use
Description: Tablet pill count
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Tablets per subject
Arm/Group | (PN 400 (VIMOVO) Twice Daily) | (Celebrex 200 mg Once Daily) | (Placebo Twice Daily)
Number analyzed (Participants) | 246 | 242 | 124
Tablets per subject | 9.3 (17.5) | 13.9 (21.6) | 15.4 (37.6)

9. Secondary Outcome: Modified Severity of Dyspepsia Assessment (mSODA)
Description: Change from Baseline in the Modified Severity of Dyspepsia Assessment (mSODA) average daily pain intensity converted total score at Week 12. The mSODA instruments consists of 6 questions about abdominal discomfort during the past 24 hours, with a converted score of 2 through 47. Lower score equals less pain.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | (PN 400 (VIMOVO) Twice Daily) | (Celebrex 200 mg Once Daily) | (Placebo Twice Daily)
Number analyzed (Participants) | 245 | 237 | 123
Scores on a scale | -3.5 (9.3) | -4.8 (9.1) | -4.0 (9.4)

10. Secondary Outcome: Percent of Days With no Heartburn (Heartburn Resolution)
Description: During 12 weeks, daily heartburn question with ratings none, mild, moderate, or severe. Percent of days with Heartburn resolution (heartburn is none).
Time Frame: 12 weeks
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: percent days
Arm/Group | (PN 400 (VIMOVO) Twice Daily) | (Celebrex 200 mg Once Daily) | (Placebo Twice Daily)
Number analyzed (Participants) | 245 | 241 | 123
percent days | 83.9 (29.8) | 75.8 (34.1) | 68.5 (37.0)

11. Secondary Outcome: Number of Participants Reporting Pre-specified Non-steroidal Antiinflammatory Drug-associated Upper Gastrointestinal (UGI) Symptoms
Description: Number of participants reporting pre-specified non-steroidal antiinflammatory drug-associated (NSAID) upper gastrointestinal (UGI) symptoms. Pre-specified NSAID-associated UGI symptoms include adverse events such as dyspepsia, abdominal pain or discomfort, nausea, vomiting.
Time Frame: daily during 12 weeks
Population: Safety population
Measure: Number; unit: participants
Arm/Group | (PN 400 (VIMOVO) Twice Daily) | (Celebrex 200 mg Once Daily) | (Placebo Twice Daily)
Number analyzed (Participants) | 247 | 243 | 124
participants | 41 | 41 | 24

12. Secondary Outcome: The Number of Subjects Who Discontinued From the Study Due to Any Pre-specified Non-steroidal Antiinflammatory Drug-associated Upper Gastrointestinal Adverse Event
Description: The number of subjects who discontinued from the study due to any pre-specified non-steroidal antiinflammatory drug (NSAID)-associated upper gastrointestinal (UGI) adverse event (as classified by MedDRA). Pre-specified NSAID-associated UGI symptoms include adverse events such as dyspepsia, abdominal pain or discomfort, nausea, vomiting.
Time Frame: daily during 12 weeks
Population: Safety population
Measure: Number; unit: participants
Arm/Group | (PN 400 (VIMOVO) Twice Daily) | (Celebrex 200 mg Once Daily) | (Placebo Twice Daily)
Number analyzed (Participants) | 247 | 243 | 124
participants | 3 | 4 | 3

ADVERSE EVENTS:
Time Frame: randomization -28 days post last dose
Arm/Group | (PN 400 (VIMOVO) Twice Daily) | (Celebrex 200 mg Once Daily) | (Placebo Twice Daily)
Serious Adverse Events (participants affected / at risk) | 5/247 | 5/243 | 0/124
Other Adverse Events (participants affected / at risk) | 118/247 | 101/243 | 77/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (PN 400 (VIMOVO) Twice Daily) (N=247) | (Celebrex 200 mg Once Daily) (N=243) | (Placebo Twice Daily) (N=124)
Appendicitis perforated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (PN 400 (VIMOVO) Twice Daily) (N=247) | (Celebrex 200 mg Once Daily) (N=243) | (Placebo Twice Daily) (N=124)
Diarrhea (Gastrointestinal disorders) | 15 (15) | 8 (8) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 13 (13) | 19 (19) | 14 (14)
Nausea (Gastrointestinal disorders) | 12 (12) | 6 (6) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 10 (10) | 9 (9) | 2 (2)
Constipation (Gastrointestinal disorders) | 9 (9) | 5 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 6 (6) | 2 (2)
Stomach discomfort (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 6 (6) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 4 (4)
Sinusitis (Infections and infestations) | 5 (5) | 3 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4) | 3 (3)
Dizziness (Nervous system disorders) | 7 (7) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 7 (7) | 10 (10) | 5 (5)
Oedema peripheral (General disorders) | 9 (9) | 3 (3) | 1 (1)
Fatigue (General disorders) | 3 (3) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No